CLINICAL TRIAL: NCT02356471
Title: Pilot Study of a Consumer-Based Activity Monitor (Fitbit Zip) in Evaluating Perioperative Activity of Older Adults Undergoing Major Oncologic Surgery
Brief Title: Consumer-Based Activity Monitor in Evaluating and Measuring Activity of Older Patients With Abdominal Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00031577; NCI-2015-00097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 02114 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-01-29; First posted 2015-02-05 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Malignant Gastrointestinal Neoplasm; Malignant Peritoneal Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive care (consumer-based activity monitor) (Experimental): Patients wear Fitbit Zip (portable pedometer device) to track physical activity for 7 days before undergoing surgery and for 21 more days after undergoing surgery.
  Interventions: Device: Management of Therapy Complications Fitbit Zip (portable pedometer device); Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Device: Management of Therapy Complications Fitbit Zip (portable pedometer device) — Use pedometer to monitor physical activity
  Other Names: complications of therapy, management of
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot clinical trial studies how well consumer-based activity monitor works in evaluating and measuring activity of older patients with abdominal cancer undergoing surgery. Consumer-based activity monitor (CAM) may identify patients who are at-risk for increased post-surgery medical problems. With early identification of at-risk patients, CAM provide supervised exercise in the preoperative and postoperative periods to improve over mobility and potentially decrease preoperative complications among patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the feasibility and adherence of using a consumer-based activity monitor during the preoperative period both in the hospital as well as at home.

SECONDARY OBJECTIVES:

I. To evaluate the ability of a consumer-based activity monitor to demonstrate a 50% decrease in average daily steps for participants before and after major oncologic surgery.

II. To characterize in-home movement among older cancer patients. III. To compare in-home CAM data to in-clinic pre- and post-operative mobility testing using the Short Physical Performance Battery (SPPB).

IV. To compare in-home CAM data to pre- and post-operative self-reported mobility using the Pepper Assessment Tool for Disability (PAT-D) and the Mobility Assessment Tool-Short Form (MAT-sf).

V. To compare in-home CAM data to self-reported daily activity data during the pre- and post-operative period.

VI. To determine estimates of future study accrual, adherence, and drop-out. VII. To obtain participant feedback from participants to determine potential study opportunities and barriers.

VIII. To identify potential key stakeholders and potential patient partners for development of future grant submissions.

IX. To summarize baseline cognitive screens, physical assessment questionnaire (Pepper Assessment Tool for Disability, PAT-D), mobility assessment tool-short form (MAT-sf), health-related quality of life (FACIT-G) questionnaire, activity questionnaire (Community Healthy Activities Model Program for Seniors [CHAMPS]), pain assessment (Pain Visual Analog Scale, PVAS), fatigue assessment (Fatigue Visual Analog Scale, FVAS), and physical function testing (Short Physical Performance Battery and time to complete 400-meter walk).

X. CAM data will be compared with research grade activity data provided by the ActiGraph.

OUTLINE:

Patients wear Fitbit Zip (portable pedometer device) to track physical activity for 7 days before undergoing surgery and for 21 more days after undergoing surgery.

After completion of study, patients are followed up at 21 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) < 3
* Histologically or cytologically confirmed gastrointestinal or peritoneal malignancy
* Scheduled for major open abdominal oncologic surgery
* Able to walk without an assistive device
* Able to complete a minimum of 4 days of in-home activity monitoring before operation
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document
* Ability to understand and complete the study survey instruments in English

Exclusion Criteria:

* Cerebrovascular accident (CVA) or stroke within the past 6 months
* Severe or symptomatic heart disease
* Currently residing in nursing or assisted living facility
* Neurologic disorder that impairs ambulation (e.g. Parkinson's)
* Actively undergoing treatment for a psychiatric illness
* Resting blood pressure > 160/100
* Clinically evident cognitive and/or behavioral impairment that in the opinion of the study investigator would impair the ability of the patient to adhere to the study procedures, specifically completing home activity monitoring
* Current alcohol or other substance abuse or history of abuse within 6 months prior to screening
* Post-operative complications that in the opinion of the study investigator would impair the ability of the patient to adhere to the study procedures, specifically completing home activity monitoring
* Unable to understand and complete the study survey instruments in English

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clancy Clark, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Started | 34
Completed | 28
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.99 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Self-report Wearing the Consumer-based Activity Monitor at Least 16 Days of the 21 Day Period
Description: Feasibility will be defined as the number of patients who self-report wearing the CAM device at least 16 days of the 21 day period.
Time Frame: 21 days
Population: 34 patients enrolled in study. 28 patients had data collected. Due to challenges associated with data collection, partial data was collected for 18 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 28
Participants | 9

2. Secondary Outcome: Change in Daily Steps for Participants Before and After Major Oncologic Surgery
Description: This outcome measure will be the change in daily steps for participants before and after major oncologic surgery. Change in median (IQR) steps reported.
Time Frame: baseline and 90 days
Population: 16 subjects had sufficient data for partial analysis.
Measure: Median (Inter-Quartile Range); unit: steps
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 16
steps | -2573 [-2685 to -2461]

3. Secondary Outcome: Change in Short Physical Performance Battery (SPPB)
Description: This outcome measure is to compare pre- and post-operative mobility using the Short Physical Performance Battery (SPPB). Median (IQR) change in SPPB from baseline to 90 days is reported.The scale range is 0-16. Higher scores denotes better outcomes.
Time Frame: baseline and 90 days
Population: Only 9 subjects had SPPB measured at baseline and 90 days.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 9
units on a scale | 0 [-1 to 2]

4. Secondary Outcome: Change in Duration of 400-meter Walk
Description: This outcome measure is to compare pre- and post-operative mobility testing using the 400-meter walk. Median (IQR) change in 400 m walk from baseline to 90 days is reported. The duration it takes the participant to walk 400 meters will be recorded in seconds.
Time Frame: baseline and 90 days
Population: Only 10 subjects had 400m walk measured at baseline and 90 days
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 10
seconds | -69.5 [-166.1 to 30.6]

5. Secondary Outcome: Change in Pepper Assessment Tool for Disability (PAT-D)
Description: This outcome measure is to compare pre- and post-operative self-reported mobility using the Pepper Assessment Tool for Disability (PAT-D). Median (IQR) change in PAT-D is reported.
Time Frame: baseline and 90 days
Population: Data were not collected and therefore analysis cannot performed.
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in the Mobility Assessment Tool-Short Form (MAT-sf).
Description: This outcome measure is to compare pre- and post-operative self-reported mobility using the Mobility Assessment Tool-Short Form (MAT-sf). Median (IQR) change in MAT-sf is reported. The score range is 30-80 and higher scores denotes better outcomes.
Time Frame: baseline and 90 days
Population: Only 7 subjects had MAT-sf measured at baseline and 90 days.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 7
units on a scale | 4.52 [-0.465 to 5.42]

7. Secondary Outcome: Change in CHAMPS Between the Pre- and Post-operative Period
Description: This outcome measure is to compare self-reported activity data (CHAMPS) during the pre- and post-operative period. Median (IQR) change in CHAMPS is reported. CHAMPS measures activity of the participant and how long they could do the activity. The score range is 0-108. Higher scores denotes better outcomes.
Time Frame: baseline and 90 days
Population: 5 subjects have CHAMPs data at baseline and 90 days.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 5
score on a scale | -1 [-1 to 2]

8. Secondary Outcome: Change in Health-related Quality of Life (FACT-G) Questionnaire
Description: FACT-G is a 27-item compilation of general questions divided into 4 primary quality of life (QOL) domains: physical well-being, social/family well-being, emotional well-being, and functional well-being. The subscales are summed to produce a total score. The total score range is 0-108 and a higher score indicates better quality of life. Outcomes is to compare FACT-G at baseline and 90 days. Change in FACT-G is reported in median (IQR).
Time Frame: baseline and 90 days
Population: Only 6 subjects reported FACT-G at baseline and 90 days.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 6
units on a scale | -1 [-1 to 2]

9. Secondary Outcome: Change in Pain Assessment -Pain Visual Analog Scale, (PVAS)
Description: The pain VAS is a unidimensional measure of pain intensity providing a range of scores from 0-100. A higher score indicates greater pain intensity. Change in median (IQR) pain score from baseline to 90 days is reported.
Time Frame: baseline and 90 days
Population: Only 6 subjects had pain VAS measured at baseline and 90 days.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 6
units on a scale | 21 [3 to 34.5]

10. Secondary Outcome: Change in Fatigue Assessment- Fatigue Visual Analog Scale (FVAS).
Description: The fatigue VAS is a unidimensional measure of fatigue providing a range of scores from 0-100. A higher score indicates greater fatigue. Change in median (IQR) fatigue score from baseline to 90 days is reported.
Time Frame: baseline and 90 days
Population: Only 6 subjects reported fatigue VAS at baseline and 90 days.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
Number analyzed (Participants) | 6
units on a scale | 6 [0 to 25.5]

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events occurred for study. Definitions used for adverse events did not differ from clinicaltrials.gov
Arm/Group | Supportive Care (Consumer-based Activity Monitor)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
This feasibility study closed early due to slow accrual and inability to capture specific study variables. Small sample size limited study analysis and prevents reliable interpretation of data collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes